CLINICAL TRIAL: NCT05065216
Title: Phase 2/3 Adaptive Design, Randomized Double-blind Placebo-controlled Study to Evaluate the Safety and Efficacy of DM199 for the Treatment of Acute Ischemic Stroke (ReMEDy2 Trial)
Brief Title: Treatment of Acute Ischemic Stroke (ReMEDy2 Trial)
Acronym: ReMEDy2
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: DiaMedica Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DM199-2021-001
Record Dates: First submitted 2021-09-03; First posted 2021-10-04 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Acute Stroke; Ischemic Stroke; Stroke
Keywords: acute; ischemic; stroke; AIS; tPA; LVO; MT; KLK1; Kallikreins
MeSH Terms: conditions — Stroke; Ischemic Stroke; Ischemia | interventions — DM199; Injections

STUDY DESIGN:
Intervention Model Description: Phase 2/3 Adaptive Design, Randomized Double-blind Placebo-controlled Study to Evaluate the Safety and Efficacy of DM199 for the Treatment of Acute Ischemic Stroke (ReMEDy2 Trial)
Who Masked: Participant, Investigator
Masking Description: To minimize bias, the participant and PI will be blinded to treatment assignment. All Sub-Investigators and other members of the study team will also remain blinded. The study team will remain blinded until all data is collected, and database lock occurs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DM199 (Experimental): DM199 administered by a single intravenous (IV) dose followed by subcutaneous (SC) doses at 2 hours (+10 hours) of the IV dose completion and then 2 times per week up to Day 21.
  Interventions: Drug: Recombinant human tissue kallikrein
- Placebo for DM199 Solution for Injection (Placebo Comparator): Placebo administered by a single intravenous (IV) dose followed by subcutaneous (SC) doses at 2 hours (+10 hours) of the IV dose completion and then 2 times per week up to Day 21.
  Interventions: Other: Placebo for DM199 Solution for Injection

INTERVENTIONS:
Drug: Recombinant human tissue kallikrein — DM199 administered by a single intravenous (IV) dose followed by subcutaneous (SC) doses at 2 hours (+10 hours) of the IV dose completion and then 2 times per week up to Day 21
  Other Names: DM199
  Arms: DM199
Other: Placebo for DM199 Solution for Injection — Placebo administered by a single intravenous (IV) dose followed by subcutaneous (SC) doses at 2 hours (+10 hours) of the IV dose completion and then 2 times per week up to Day 21.
  Arms: Placebo for DM199 Solution for Injection

SUMMARY:
This is a Phase 2/3 study evaluating the safety and efficacy of DM199 (rinvecalinase alfa) in treating participants with moderate stroke severity, who present within 24 hours of Acute Ischemic Stroke (AIS) onset due to small and medium vessel occlusions. This study focuses on participants with limited treatment options. Participants who have or will receive mechanical thrombectomy (MT) are not eligible for participation. Additionally, participants who have received fibrinolytics are excluded unless they experience a persistent neurological deficit of moderate severity six or more hours after fibrinolytic treatment. Participants considered for this trial should not be denied the use of standard of care (SoC) AIS therapies, such as fibrinolytics or MT, when appropriate. The double-blinded study will be randomized and placebo-controlled at up to approximately 100 sites.

DETAILED DESCRIPTION:
This is a Phase 2/3 Adaptive Design, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of DM199 for the Treatment of Acute Ischemic Stroke (ReMEDy2 Trial). Participants with AIS will be randomized 1:1 to DM199 or placebo. DM199 will be administered as a single intravenous (IV) dose (0.5 μg/kg; not to exceed 50 μg) followed by subcutaneous (SC) doses at 2 hours (+10 hours) of the IV dose completion and then 2 times per week up to Day 21. The duration of each individual's participation in the study will be approximately 90 days from the time of initial treatment to completion of all study activities.

A formal interim analysis will be conducted after 200 participants complete their Day 90 assessment in Part A. The purposes of this interim analysis are to assess safety, allow early stopping of the study for futility, or continuing the study with a revised final sample up to a maximum of 728 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is between 18 and 90 years of age inclusive.
2. Participant weight is 40 kg to 166 kg inclusive.
3. Participant to be randomized and treatment initiated within 24 hours of last known normal/AIS stroke onset.
4. Participant has NIHSS ≥5 and ≤15 at approximately the time of randomization. This criterion also applies to participants who meet the following conditions:

   * The participant initially presents with an NIHSS score below 5 but clinically worsens, including cases of progressing stroke / stroke-in-evolution, resulting in a subsequent persistent NIHSS score of ≥5 and ≤15; and
   * Participant meets all other inclusion and exclusion criteria, including repeat brain imaging to rule out hemorrhagic transformation.
5. Participant had a pre-morbid mRS score of 0 to 1 (mRS score prior to AIS) as stated by participant or participant's representative.
6. If participant has received fibrinolytic treatment for AIS within 4.5 hours of last know normal/AIS stoke onset and at least 6 hours after completing fibrinolytic treatment, and the participant meets all of the following criteria:

   * Participant's initial NIHSS score prior to fibrinolytics was ≤15; and
   * At least six hours after fibrinolytics, the participant has NIHSS score of ≥5 and ≤15 with a persistent deficit; and
   * The participant's NIHSS score showed less than a 4-point improvement, or worsened, after receiving fibrinolytics; and
   * Participant meets all other inclusion and exclusion criteria including repeat brain imaging to rule out hemorrhagic transformation.
7. Participant and/or legally authorized representative is able to provide informed consent.
8. Participant is willing and able to comply with the study protocol, in the Investigator's judgment.

Exclusion Criteria:

1. At screening, or with repeat imaging (see Inclusion 4 and 6), participant has imaging confirmed hemorrhage stroke.
2. Participant has image findings with symptomatic large vessel occlusion at one or more of the following locations: Intracranial carotid I/T/L or M1 segment MCA, vertebral or basilar artery (BA).
3. Participant has large core of established infarction defined as ASPECTS 0-5.
4. Participant has or will receive MT for their current AIS.
5. Participant has suspected or confirmed extracranial arterial dissection.
6. Participant has imaging findings and/or symptoms consistent with a brain stem or cerebellar stroke. Posterior cerebral artery strokes without any associated brain stem or cerebellar involvement are allowable.
7. Participant has any recorded SBP <100 mmHg or MAP <65 mmHg; MAP = DBP + [1/3 (SBP - DBP)] (measured with noninvasive BP cuff type monitor) after stroke symptom onset and prior to randomization.
8. Participant is currently prescribed angiotensin-converting enzyme inhibitor (ACEi) and is unable or unwilling to convert to another antihypertensive pharmacological treatment through Day 29 ±1 day (8 days after last treatment).
9. Participant is currently prescribed an ACEi, and the last dose of the ACE inhibitor medication is reported to have been taken < 24 hours before start of IV study drug infusion as stated by participant or participant's representative.
10. Participant has a history of clinically significant allergic reactions such as angioedema or anaphylaxis requiring hospitalization.
11. Participant has a diagnosis or suspected diagnosis of hereditary angioedema (HAE) or is taking or prescribed medications commonly used as prophylaxis/treatment of HAE, such as C1-esterase inhibitors (Cinryze, Berinert, Ruconest, Haegarda), Danazol, kallikrein inhibitors (Ecallantide, Berotralstat, Lanadelumab), Bradykinin B2 Receptor Antagonists (Icatibant), or other medication designed to influence the kallikrein-kinin system.
12. Life expectancy estimated at ≤1 year prior to enrollment.
13. Participant has clinical evidence of an active infection at the time of enrollment requiring parenteral treatment or hospitalization to monitor or manage the infection.

    NOTE: Treatment of uncomplicated infections with oral antibiotics would not be an exclusion (for example, the treatment of uncomplicated urinary tract infections or sinus infections with oral antibiotics would not be exclusionary).
14. Participant has known alpha 1-antitrypsin deficiency (α1-antitrypsin deficiency).
15. Participant is pregnant or nursing. NOTE: Participants who agree to stop nursing may be considered for inclusion at the discretion of the Investigator.
16. Participants of child-bearing potential must agree to use medically acceptable contraceptive measures to prevent pregnancy. All participants of childbearing potential (defined as sexually mature participants who have had menses within the preceding 24 months and have not undergone permanent sterilization methods such as hysterectomy, bilateral oophorectomy, bilateral salpingectomy, etc.) must have a negative serum pregnancy test performed locally at screening. Participants of childbearing potential must agree not to attempt to become pregnant or undergo in vitro fertilization. If participating in sexual activity that could lead to pregnancy, participants must use 2 reliable methods (1 per partner is acceptable) of contraception simultaneously while receiving protocol-specified medication and during the study follow-up period.

    Participants participating in sexual activity must agree to use, or for their partner to use highly effective birth control methods (those with a failure rate of less than 1% per year when used consistently and correctly) until they have completed the study (after the Day 90 visit). Such methods include:
    * Combined (estrogen and progesterone containing) hormonal oral, intravaginal, or transdermal contraception associated with the inhibition of ovulation
    * Progesterone-only oral, injectable, or implantable hormonal contraception associated with the inhibition of ovulation
    * Intrauterine device (IUD)
    * Intrauterine hormone-releasing system (IUS)
    * Bilateral tubal occlusion
    * Vasectomized partner
    * Sexual abstinence Participants who are not of reproductive potential (who have been postmenopausal for more than 24 consecutive months or have undergone hysterectomy, bilateral oophorectomy, bilateral salpingectomy, etc.) are not required to use contraception.

    Participants are prohibited from sperm donation. NOTE: A negative serum pregnancy test will be documented during screening if a participant is of child-bearing potential.
17. Participant is currently participating in or has participated in a study using an investigational device or drug or received an investigational drug or investigational use of a licensed drug within 30 days prior to screening.
18. Participant does not have sufficient venous access for infusion of study treatment or blood sampling.
19. Participant is unable or unwilling to comply with protocol requirements, including assessments, tests, and follow-up visits.
20. Participant has any other medical condition which in the opinion of the Investigator will make participation medically unsafe or interfere with the study results.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 728 (Estimated)
Dates: Start 2021-11-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Stroke Recovery | Day 90
  Stroke recovery as defined by participants with excellent functional outcomes at Day 90 as assessed via the Modified Rankin Score (mRS [dichotomized]), mRS scores of 0 or 1 represent responders, scale range of 0-6.
  The mRS (Modified Rankin Scale) is a single-item, clinician-reported measure of functional disability in participants with AIS. Scores range in grade from 0 (no symptoms at all) to 6 (participant death).

SECONDARY OUTCOMES:
Effect on Disability | Day 90
  Assessment of effect on disability across the full spectrum of AIS by examining the distribution of mRS (shift) scores (scale range = 0 to 6) at Day 90. The mRS (Modified Rankin Scale) is a single-item, clinician-reported measure of functional disability in participants with AIS. Scores range in grade from 0 (no symptoms at all) to 6 (participant death).
Independent Function | Day 90
  Proportion of participants achieving independent function (able to look after their own affairs without assistance) with or without minor disability at Day 90 assessed as mRS 0-2 (dichotomized) mRS scores of 0, 1 or 2 represent responders, scale range of 0-6. The mRS (Modified Rankin Scale) is a single-item, clinician-reported measure of functional disability in participants with AIS. Scores range in grade from 0 (no symptoms at all) to 6 (participant death).
Mortality Rate | Day 90
  Mortality rate as defined by event rate (%) for mortality over 90 days.
Neurological Outcome | Day 90
  Proportion of participants achieving an excellent neurological outcome defined by National Institute of Health Stroke Scale (NIHSS)= 0-1 (dichotomized) (NIHSS scores of 0 or 1, scale range 0 to 42) at Day 90.
  The National Institute of Health Stroke Scale (NIHSS) is a clinician-reported measure used to rate the severity of strokes, namely disability and recovery after acute stroke. The scale is comprised of 11 items with item scores ranging from 0 to 4. Total scores range from 0 to 42, with higher scores indicating increased severity.
Functional Independence | Day 90
  Proportion of participants achieving an excellent functional independence in activities of daily living defined by Barthel Index score (dichotomized) greater than or equal to 5 (scale range 0 to 100) at Day 90.
  The Barthel Index (BI) is a 10-item scale assessing activities of daily living and functional disability. Each item is scored in increments of 5 points (0, 5, 10, or 15) and the individual items are summed to produce a total score between 0 and 100, with higher scores representing more optimal performance (100 = fully independent) and lower scores representing inferior performance (0 = totally dependent).
AIS Recurrence | Day 90
  Recurrent AIS as defined by proportion of participants who experience a recurrent AIS by Day 90 as assessed by a new, persistent neurological deficit attributable to cerebrovascular ischemia. Imaging findings, if available, should support the diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Volpi, M.D., Principal Investigator — The Methodist Hospital Research Institute; Rachel Laursen, M.D., Principal Investigator — Oregon Health & Science University (OHSU)
Locations (42):
- United States (32):
  - Gulf Health Hospitals d/b/a Thomas Hospital, Fairhope, Alabama
  - USC Arcadia Hospital, Arcadia, California
  - Glendale Adventist Medical Center d/b/a Adventist Health Glendale, Glendale, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - The Lundquist Institute at Harbor UCLA Medical Center, Torrance, California
  - Memorialcare Long Beach Medical Center, Torrance, California
  - HCA Florida - JFK Medical Center, Atlantis, Florida
  - University of Florida Jacksonville, Jacksonville, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Tampa General Hospital (TGH) - The Stroke Center, Tampa, Florida
  - OSF HealthCare Saint Francis Medical Center, Peoria, Illinois
  - Community Hospital - MacArthur, Munster, Indiana
  - Ascension Via Christi Hospitals Wichita Inc., Wichita, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - UMASS Chan Medical School, Worcester, Massachusetts
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - The University of New Mexico - School of Medicine, Albuquerque, New Mexico
  - Northwell Health Physician Partners - Neurology at Lenox Hill, New York, New York
  - Summa Health Clinical Research Center, Akron, Ohio
  - The Clinical Neuroscience Institute, Dayton, Ohio
  - Mercy Health - St. Vincent Medical Center, Toledo, Ohio
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Ascension St. John, Tulsa, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Prisma Health-Greenville Memorial Hospital, Greenville, South Carolina
  - Erlanger Hospital, Chattanooga, Tennessee
  - Chattanooga Center for Neurologic Research, Chattanooga, Tennessee
  - Houston Methodist Neurological Institute, Houston, Texas
  - Memorial Hermann Hospital, Texas Medical Center, Houston, Texas
- Canada (4):
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Health Sciences North, Hamilton, Ontario
  - Hamilton Health Sciences - Hamilton General Hospital, Hamilton, Ontario
- Georgia (5):
  - West Georgia Medical Center LTD, Kutaisi, Georgia
  - Israel-Georgia Medical Research Clinic-Healthycore LTD, Tbilisi, Georgia
  - New Hospitals LTD, Tbilisi, Georgia
  - Pineo Medical Ecosystem LTD, Tbilisi, Georgia
  - JSC K. Eristavi National Center of Experimental and Clinical Surgery, Tbilisi, Georgia
- Royal Stoke University Hospital, Stoke-on-Trent, United Kingdom, United Kingdom

IPD SHARING:
Plan to Share IPD: No